CLINICAL TRIAL: NCT06983756
Title: " Evaluation of Erythropoietin Therapy in Patients With End-Stage Kidney Disease on Regular Hemodialysis: Hemoglobin Outcomes, and Metabolic Syndrome as a Risk Factor for Erythropoietin Resistance "
Status: Not yet recruiting | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nada Elsayed Abdeltwab Issa, Teaching Assistant, Fayoum University
Other Study IDs: Erythropoietin Resistance & MS
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Erythropoietin Resistant Anemia (EPO Resistant Anemia)
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: participants with metabolic syndrome
  Interventions: Drug: Erythropoietin
- group 2: participants without metabolic syndrome
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — EPO resistance

SUMMARY:
The primary aim of this study is to investigate the association between metabolic syndrome and erythropoietin resistance in patients with End-Stage Kidney Disease (ESKD).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a common condition that has significant implications for patients' health and healthcare budgets. CKD is a major contributor to morbidity and mortality across the globe. The incidence and prevalence of CKD are rising steadily all over the world. Along with many adverse effects on different body organs, CKD and end-stage kidney disease (ESKD) are associated with body will beting and malnutrition. Patients with ESKD require maintenance hemodialysis (MHD) to sustain their life.

Patients with chronic kidney disease (CKD) have a relatively deficient erythropoietin (EPO) production, and this is the main cause of anemia in this group. In its severe form, anemia decreases quality of life and increases the risk of cardiovascular diseases and mortality in dialysis patients, so the implementation of prevention and control measures is recommended [4]. Erythropoiesis-stimulating agents (ESAs) are generally used to control anemia and reduce the need for blood transfusions in patients with CKD.

ESA resistance or hyporesponsiveness occurs when the patient does not reach the desired serum hemoglobin (Hb) concentration even with the use of ESA at doses higher than usual or when increasingly higher doses are necessary to maintain the recommended Hb concentration.

The main causes of EPO resistance are iron deficiency, chronic inflammation, inadequate dialysis, hyperparathyroidism, hemolysis, vitamin B12, and folate deficiency. Observational studies have shown that nutritional status is associated with EPO resistance in HD patients, mainly because of malnutrition-inflammation status.

While treating anemic patients with αEPO can increase hemoglobin levels to recommended values and decrease complications in hemodialysis patients, the treatment of anemia with an ESA can increase the risk of mortality; high dosages of the ESA and treatment resistance are the primary factors for this outcome. Thus, it is important to determine which factors limit the ability of αEPO to correct anemia in hemodialysis patients so that treatment can be optimized.

ELIGIBILITY:
Inclusion Criteria:

* Patients (and replacements) will be randomly selected by a raffle.
* All participants should be 18 years of age or older and agree to participate in the study after due clarification.
* Patients with end stage kidney disease (ESKD) on regular hemodialysis for more than 3 months.

Exclusion Criteria:

* - Patients with neoplasm, severe cardiovascular, cerebrovascular and liver diseases.
* Females with polycystic ovarian syndrome, those on hormonal replacement therapy and pregnant women.
* Patients with infection or autoimmune diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients who will be enrolled in this study are receiving recombinant human erythropoietin therapy with epoetin alfa (αEPO), used to control anemia at our reference hospital.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
HB | 6 month
  Hemoglobin in blood

REFERENCES:
- [Background] Carney EF. The impact of chronic kidney disease on global health. Nat Rev Nephrol. 2020 May;16(5):251. doi: 10.1038/s41581-020-0268-7. No abstract available. PMID 32144399
- [Background] Eriguchi R, Taniguchi M, Ninomiya T, Hirakata H, Fujimi S, Tsuruya K, Kitazono T. Hyporesponsiveness to erythropoiesis-stimulating agent as a prognostic factor in Japanese hemodialysis patients: the Q-Cohort study. J Nephrol. 2015 Apr;28(2):217-25. doi: 10.1007/s40620-014-0121-9. Epub 2014 Jul 31. PMID 25080399